CLINICAL TRIAL: NCT02728739
Title: Incidence of Significant Mitral Regurgitation in Patients Presenting With Acute Heart Failure: Journey to Tertiary Centre
Brief Title: Incidence of Significant Mitral Regurgitation in Acute Heart Failure Patients
Acronym: MRAHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metanoic Health Ltd. (Industry)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHL-2016-001
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Acute Heart Failure; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute Heart Failure Patients (Experimental): Acute Heart Failure patients with elevated levels of BNP ( >30pg/ml) will undergo Transthoracic Echocardiogram (TTE) for grading of MR severity within 7 days.
  Interventions: Procedure: Transthoracic Echocardiogram (TTE) Assesment

INTERVENTIONS:
Procedure: Transthoracic Echocardiogram (TTE) Assesment — Transthoracic Echocardiogram (TTE) will be carried out on all heart failure patients with elevated BNP level (>30 pg/ ml) for grading of MR severity within 7 days.

SUMMARY:
The purpose of this study is to determine the prevalence of moderate-to-severe Mitral Regurgitation (MR) in acute Heart Failure (HF) patients requiring hospital admission.

DETAILED DESCRIPTION:
All patients admitted with symptoms of HF- (shortness of breath (SOB), peripheral oedema, palpitations and irregular heart beats) will be assessed by the Research Team. The level of BNP will be checked using a small device (i-STAT BNP) at the bedside. If results of the test suggest HF they will undergo special procedure called transthoracic echocardiography (TTE). TTE is an ultrasound scan of the heart which will enable the investigators' to grade severity of Mitral Regurgitation (MR) as well as strength of the heart muscle. The investigators will use bi-plane Simpton's method to calculate left ventricular (LV) ejection fraction (EF). Colour Doppler and PISA method will be used to quantify severity of MR or valve leak. Simultaneously there will be recording of heart sounds to find out if auscultation is reliable in identifying leaky valves.

ELIGIBILITY:
Inclusion Criteria:

* Acute Heart Failure patients admitted to the Hospital
* Elevated BNP level (>30pg/ml)

Exclusion Criteria:

* Patients with BNP level (< 30pg/ml)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Grade 3 and above mitral regurgitation in acute heart failure. | 12 months
  TTE Grading is done on colour Doppler and proximal isovelocity surface area (PISA) method.

SECONDARY OUTCOMES:
Establish correlation between BNP level and severity of MR in acute HF | 12 months
  Standard statistical analysis of BNP level and grade of MR severity
The validity of Hospital Episode Statistics (HES) data against prevalence of grade 3-4 MR in the study. | 12 month
  Standard statistical analysis of 2 sets of data

CONTACTS AND LOCATIONS:
Overall Officials: Aigul Baltabaeva, MBBS MD PhD, Principal Investigator — Ashford & St Peter's Hospitals NHS Foundation Trust
Locations (1):
- St Peter's Hospital, Guildford Road, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Bonis M, Maisano F, La Canna G, Alfieri O. Treatment and management of mitral regurgitation. Nat Rev Cardiol. 2011 Nov 22;9(3):133-46. doi: 10.1038/nrcardio.2011.169. PMID 22105677
- [Background] Enriquez-Sarano M, Sundt TM 3rd. Early surgery is recommended for mitral regurgitation. Circulation. 2010 Feb 16;121(6):804-11; discussion 812. doi: 10.1161/CIRCULATIONAHA.109.868083. No abstract available. PMID 20159841
- [Background] Enriquez-Sarano M, Avierinos JF, Messika-Zeitoun D, Detaint D, Capps M, Nkomo V, Scott C, Schaff HV, Tajik AJ. Quantitative determinants of the outcome of asymptomatic mitral regurgitation. N Engl J Med. 2005 Mar 3;352(9):875-83. doi: 10.1056/NEJMoa041451. PMID 15745978
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Derived] Berrill M, Beeton I, Fluck D, John I, Lazariashvili O, Stewart J, Ashcroft E, Belsey J, Sharma P, Baltabaeva A. Disproportionate Mitral Regurgitation Determines Survival in Acute Heart Failure. Front Cardiovasc Med. 2021 Dec 2;8:742224. doi: 10.3389/fcvm.2021.742224. eCollection 2021. PMID 34926604